CLINICAL TRIAL: NCT00041249
Title: Efficacy And Safety Study Of Brostallicin In Patients With Locally Advanced Or Metastatic Soft Tissue Sarcoma Failing One Prior Chemotherapy Treatment
Brief Title: Brostallicin in Treating Patients With Locally Advanced or Metastatic Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-62011; EORTC-62011
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Gastrointestinal Stromal Tumor; Sarcoma
Keywords: adult angiosarcoma; adult fibrosarcoma; adult leiomyosarcoma; adult liposarcoma; adult neurofibrosarcoma; adult synovial sarcoma; stage III adult soft tissue sarcoma; recurrent adult soft tissue sarcoma; adult malignant fibrous histiocytoma; adult malignant hemangiopericytoma; adult rhabdomyosarcoma; gastrointestinal stromal tumor; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Sarcoma; Hemangiosarcoma; Fibrosarcoma; Leiomyosarcoma; Liposarcoma; Neurofibrosarcoma; Sarcoma, Synovial; Histiocytoma, Malignant Fibrous; Hemangiopericytoma, Malignant; Rhabdomyosarcoma | interventions — brostallicin

INTERVENTIONS:
Drug: brostallicin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of brostallicin in treating patients who have locally advanced or metastatic soft tissue sarcoma that has not responded to one previous chemotherapy regimen.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of brostallicin, in terms of objective response, in patients with locally advanced or metastatic soft tissue sarcoma who have failed one prior chemotherapy treatment.
* Determine the time to progression and duration of response in patients treated with this drug.
* Determine the safety and toxic effects of this drug in these patients.
* Correlate clinical outcome with whole blood glutathione level in patients treated with this drug.

OUTLINE: This is a multicenter study. Patients are stratified according to tumor (tumors other than gastrointestinal stromal tumor (GIST) vs GIST).

Patients receive brostallicin IV over 10 minutes on day 1. Treatment repeats every 21 days for at least 4 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 months for 1 year and then every 4 months for 1 year.

PROJECTED ACCRUAL: A total of 58-72 patients (40 for stratum I and 18-32 for stratum II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed soft tissue sarcoma that is not amenable to surgery, radiotherapy, or combined modality therapy with curative intent
* Stratum I

  * Malignant fibrous histiocytoma
  * Liposarcoma
  * Rhabdomyosarcoma
  * Synovial sarcoma
  * Malignant paraganglioma
  * Fibrosarcoma
  * Leiomyosarcoma
  * Angiosarcoma including hemangiopericytoma
  * Malignant peripheral nerve sheath tumor
  * Unclassified sarcoma
  * Miscellaneous sarcoma
* Stratum II

  * Gastrointestinal stromal tumor
  * Previously treated with imatinib mesylate for locally advanced or metastatic disease and demonstrated disease progression
* The following sarcoma types are excluded:

  * Mixed mesodermal tumors of the uterus (and carcinosarcoma)
  * Chondrosarcoma
  * Malignant mesothelioma
  * Neuroblastoma
  * Osteosarcoma
  * Ewing's sarcoma
  * Embryonal rhabdomyosarcoma
* At least one measurable lesion
* Progressive disease after 1 prior anthracycline- and/or alkylating-containing chemotherapy regimen for locally advanced or metastatic disease
* Clinical evidence of progression within 6 weeks prior to study treatment
* No known or symptomatic CNS metastases

PATIENT CHARACTERISTICS:

Age:

* Over 15

Performance status:

* WHO 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 4,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.25 times upper limit of normal (ULN)
* SGPT and SGOT no greater than 3 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 1.4 mg/dL OR
* Creatinine clearance greater than 65 mL/min

Cardiovascular:

* No prior severe cardiovascular disease

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception during and for up to 6 months after study
* No other prior or concurrent malignancy except adequately treated basal cell skin cancer or carcinoma in situ of the cervix
* No other severe medical illness
* No psychosis

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent biologic response modifiers or immunotherapy
* No concurrent prophylactic hematopoietic growth factors (e.g., filgrastim (G- CSF) or sargramostim (GM-CSF)

Chemotherapy:

* See Disease Characteristics
* More than 4 weeks since prior chemotherapy and recovered
* Prior adjuvant chemotherapy as first-line treatment allowed provided disease progressed within 6 months after the completion of chemotherapy
* No prior ecteinascidin 743 (stratum I)
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy

Radiotherapy:

* See Disease Characteristics
* Recovered from prior radiotherapy
* No prior radiotherapy to sole measurable lesion
* Concurrent palliative radiotherapy to nontarget lesions allowed at investigator's discretion

Surgery:

* See Disease Characteristics
* Recovered from prior surgery

Other:

* No other concurrent anticancer therapy (approved or investigational)
* No concurrent participation in any other clinical treatment study
* No other concurrent investigational drugs

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2002-05; Primary Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Leahy, MBChB, FRACP, FRCP, FRC Path, Study Chair — Fremantle Hospital
Locations (16):
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
- France (3):
  - Centre Leon Berard, Lyon
  - CHU de la Timone, Marseille
  - Institut Gustave Roussy, Villejuif
- Germany (4):
  - Robert Roessle Klinik, Berlin
  - Universitaets-Krankenhaus Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum Grosshadern der Ludwig-Maximilians Universitaet Muenchen, Munich
- Netherlands (4):
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam
  - Academisch Ziekenhuis Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Daniel Den Hoed Cancer Center at Erasmus University Medical Center, Rotterdam
- United Kingdom (3):
  - St. James's University Hospital, Leeds, England
  - Royal Marsden NHS Trust - London, London, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England

REFERENCES:
- [Result] Leahy M, Ray-Coquard I, Verweij J, Le Cesne A, Duffaud F, Hogendoorn PC, Fowst C, de Balincourt C, di Paola ED, van Glabbeke M, Judson I, Blay JY; European Organisation for Research and Treatment of Cancer Soft Tissue and Bone Sarcoma Group. Brostallicin, an agent with potential activity in metastatic soft tissue sarcoma: a phase II study from the European Organisation for Research and Treatment of Cancer Soft Tissue and Bone Sarcoma Group. Eur J Cancer. 2007 Jan;43(2):308-15. doi: 10.1016/j.ejca.2006.09.014. Epub 2006 Nov 13. PMID 17095209
- [Result] Leahy MG, Blay JY, Verweij J, et al.: EORTC 62011: phase II trial of brostallicin for soft tissue sarcoma. [Abstract] Eur J Cancer Suppl 1 (5): S209, A-694, 2003.